CLINICAL TRIAL: NCT05119556
Title: Video Telehealth Pulmonary Rehabilitation to Reduce Hospital Readmission in Chronic Obstructive Pulmonary Disease (Tele-COPD)
Brief Title: Video Telehealth Pulmonary Rehabilitation to Reduce Hospital Readmission in Chronic Obstructive Pulmonary Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Surya P Bhatt, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300008210; 1UG3HL155806-01A1 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2021-11-15 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Pulmonary Rehabilitation; Telehealth
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This is a 52 week, prospective, randomized controlled, phase 3, multi-center clinical trial.
Who Masked: Outcomes Assessor
Masking Description: A blinded adjudication committee will evaluate all hospitalizations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Participants will receive standard of care for COPD management per local guidance. In addition, they will receive 4-weekly phone calls for 13 weeks post discharge to inquire about health status and exacerbations.
- Video Telehealth Pulmonary Rehabilitation (Active Comparator): In addition to standard of care, participants will be asked to participate in rehabilitation sessions administered at home via live videoconferencing for approximately 60 minutes a session, three times a week. A total of 36 sessions will be planned to be completed by week 13 post-discharge. Exacerbations and health status will be ascertained every 4-weeks for 13 weeks.
  Interventions: Behavioral: Video Telehealth Pulmonary Rehabilitation

INTERVENTIONS:
Behavioral: Video Telehealth Pulmonary Rehabilitation — Participant will be asked to exercise 3 times a week at their home for 60 minutes each session, via live two-way videoconferencing using a data-enabled smart phone or similar device. A total of 36 sessions will be administered over 13 weeks post-discharge. Sessions will be administered by exercise physiologists located at the University of Alabama at Birmingham. Each session will be scheduled with up to three other participants at a time to mimic group sessions as delivered at center-based pulmonary rehabilitation programs. Exercise sessions will include aerobics, strength or resistance training, breathing exercises, and education sessions. The exercise plans will be tailored according to the participants' baseline exercise tolerance as determined by an initial six minute walk test and their answers to the questionnaires at the baseline visit.
  Arms: Video Telehealth Pulmonary Rehabilitation

SUMMARY:
The purpose of this study is to compare the efficacy and safety of a real time video telehealth pulmonary rehabilitation intervention with standard of care in patients hospitalized for an exacerbation of chronic obstructive pulmonary disease (COPD) to determine the impact on hospital readmissions and respiratory morbidity, and to investigate the cost-effectiveness of the intervention.

DETAILED DESCRIPTION:
This is a 52 week, prospective, randomized controlled, phase 3, multi-center clinical trial (n=768 at 14 clinical sites) comparing the efficacy and safety of a real time video telehealth pulmonary rehabilitation intervention with standard of care in patients hospitalized for COPD exacerbation to determine the impact on hospital readmissions and respiratory morbidity, and to investigate the cost-effectiveness of the intervention.

All patients with a clinical diagnosis of COPD who are hospitalized for an acute exacerbation of COPD at each clinical site will be considered for inclusion. Interested participants will be seen at 8 (-3 to +4) days after discharge from the hospital. At this visit, participants will be randomized 1:1, in varying blocks, stratified by site, to video telehealth PR plus standard of care versus standard of care alone. The telehealth intervention will involve 3 exercise sessions a week for 12 weeks. Exercise sessions will be provided in real-time via live two-way videoconferencing using a HIPAA-compliant app on an encrypted smart phone or similar device. Each session will be standardized to include cardiovascular (aerobic) training, strength (resistance) training, breathing exercises, and education that includes smoking cessation counselling where applicable, inhaler use techniques, diet, and nutrition. Participants in both the intervention and control arms will receive standard of care per local guidance. During the period of active intervention, participants in both arms will be contacted monthly to ascertain any exacerbations. Questionnaires and assessments of function will be administered at the baseline 8 day visit and at completion of the intervention at 13 weeks. Subsequently, participants in both arms will be called 3-monthly to ascertain healthcare utilization, and questionnaires and assessments of function will be repeated at the end of the follow-up period at 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 or greater
2. Clinical diagnosis of COPD
3. Hospitalized for acute exacerbation of COPD.
4. Be willing to adhere to trial and follow-up procedures and give informed consent

Exclusion Criteria:

1. Secondary diagnosis of congestive heart failure that is severe as documented by active symptoms, New York Heart Association (NYHA) functional classification IV or left ventricular ejection fraction <25% on echocardiography
2. Other respiratory conditions that could confound the diagnosis such as asthma, pulmonary fibrosis, bronchiectasis, and lung cancer. Participants with pneumonic exacerbations of COPD will be included.
3. Primary diagnosis of COVID pneumonia. Individuals with incidentally detected COVID or persistently positive for COVID but deemed to be convalescent will not be excluded.
4. Active cancers on chemotherapy or radiation therapy
5. Immunosuppressed states predisposing to frequent hospitalizations including uncontrolled HIV/AIDS
6. Active or recent (within 1 month) myocardial infarction
7. Angina not well-controlled by medication
8. Unstable cardiac arrhythmias, atrial or ventricular
9. Supplemental oxygen requirement greater than 5 liters per minute at either rest or with exertion
10. Significant cognitive dysfunction, including dementia, that in opinion of investigator would impair ability to safely or effectively engage in study protocol
11. Participants with any terminal medical illnesses as diagnosed by a physician, and/or on hospice
12. Currently enrolled in and participating in pulmonary rehabilitation
13. Treatment with chronic or newly initiated home ventilatory support. Those on in-patient short-term non-invasive ventilation will not be excluded.
14. Special patient groups such as prisoners and institutionalized patients
15. Participants with musculoskeletal comorbidities or physical infirmities that preclude participation in an exercise program
16. Current participation in any other interventional clinical trial
17. Inability to understand and speak English during exercise sessions
18. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
All-cause hospitalization within 30 days post discharge for an index admission for COPD exacerbation | 30 days
  Hospitalizations will be ascertained via weekly phone calls. Hospitalization for any reason will be considered a primary event when it occurs within the first 30 days after index hospitalization.
Change in St. George's Respiratory Questionnaire | 13 weeks
  The St. George's Respiratory Questionnaire (SGRQ) is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. It consists of 40 questions, and scores range from 0 to 100, with higher scores indicating worse quality of life. The minimum clinically important difference (MCID) is 4 units.
Change in six-minute walk distance | 13 weeks
  The six-minute walk test is an assessment of functional capacity, and is the distance walked in 6 minutes. The minimum clinically important difference (MCID) for COPD is 26 m.
Change in the University of California, San Diego Shortness of Breath Questionnaire | 13 weeks
  The University of California, San Diego Shortness of Breath Questionnaire (SOBQ) is a 24-question, self-administered questionnaire which rates dyspnea associated with activities of daily living. Scores range from 0 to 120, with higher scores indicating greater dyspnea. The minimum clinically important difference (MCID) is 5.
Cost Savings | 30 days
  Cost saving will be estimated by comparing costs of the intervention and savings resulting from readmission reduction within 30 days.
Cost per Quality Adjusted Life Year Gained | 52 weeks
  Cost-effectiveness will be calculated by comparing Telehealth PR with Standard of Care using incremental cost-effectiveness ratios.

SECONDARY OUTCOMES:
90-days all cause readmission rate | 13 weeks
  Hospitalizations will be ascertained by healthcare utilization questionnaire at the weekly phone calls.
The adverse events (AEs) and serious adverse events (SAEs) | 13 weeks
  Safety of video telehealth PR intervention as determined by adverse events (AEs) and serious adverse events (SAEs)
Change in COPD Assessment Test score | 13 weeks
  The COPD Assessment Test (CAT) survey is a validated, short (8-item) and simple patient completed questionnaire, and measures the health status of patients with COPD. This score is responsive to interventions such as pulmonary rehabilitation with a minimum clinically important difference (MCID) of 2 units.
Change in 30-second Sit-to-Stand Test | 13 weeks
  The 30-second Sit-to-Stand test is an assessment of skeletal muscle dysfunction, leg strength and endurance. Scores range from 4 to 14, depending on age and sex, and higher scores indicate higher levels of functioning. The minimum clinically important difference (MCID) is 2.
Change in the Clinical visit-PROactive Physical Activity Score | 13 weeks
  The Clinical visit-PROactive Physical Activity in COPD (C-PPAC) questionnaire will be used to generate scores for amount of physical activity, difficulty with physical activity and total physical activity experience. C-PPAC scores will be calculated by combining questionnaire items with two variables from activity monitors (steps/day and vector magnitude units (VMU)/min). Scores range from 0 to 100, where higher numbers indicate a better score. The minimum clinically important difference (MCID) is 6 for the amount and difficulty scores and 4 for the total score.
Change in Pulmonary Rehabilitation Adapted Index of Self-Efficacy | 13 weeks
  The Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE) tool is a 15-item disease-specific questionnaire that measures pulmonary rehabilitation-specific self-efficacy. The score ranges from 15 to 60, with higher scores indicating high levels of self-efficacy. The minimum clinically important difference (MCID) is 1.5 units.
Change in Pittsburgh Sleep Quality Index | 13 weeks
  The Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality over a 1-month time interval. It has 7 components (sleep quality, latency, duration, efficiency, disturbance, medication use, and daytime dysfunction) that are each scored from 0 to 3 for a total PSQI score of 0 to 21, with higher scores indicating worse sleep quality. The minimum clinically important difference (MCID) is 3 units.
Change in Hospital Anxiety and Depression Scale | 13 weeks
  The Hospital Anxiety and Depression Scale (HADS) will be used to measure symptoms of anxiety and depression. The HADS contains 14 items and consists of two subscales: anxiety and depression. Each item is rated on a four-point scale, with maximum scores of 21 for anxiety and depression. The minimum clinically important difference (MCID) is 1.5 units.
Change in The modified Medical Research Council score | 13 weeks
  The modified Medical Research Council (mMRC) has 5 questions that assess dyspnea in a graded fashion and quantify symptoms in COPD. The minimum clinically important difference (MCID) is 0.7.

OTHER OUTCOMES:
12-month all-cause hospitalizations | 52 weeks
  Hospitalizations following the index admission will be ascertained by healthcare utilization questionnaire at the weekly and monthly phone calls.
Change in COPD Assessment Test score | 52 weeks
  The COPD Assessment Test (CAT) survey is a validated, short (8-item) and simple patient completed questionnaire, and measures the health status of patients with COPD. This score is responsive to interventions such as pulmonary rehabilitation with a minimum clinically important difference (MCID) of 2 units.
Change in 30-second Sit-to-Stand Test | 52 weeks
  The 30-second Sit-to-Stand test is an assessment of skeletal muscle dysfunction, leg strength and endurance. Scores range from 4 to 14, depending on age and sex, and higher scores indicate higher levels of functioning. The minimum clinically important difference (MCID) is 2.
Change in Clinical visit-PROactive Physical Activity Score | 52 weeks
  The Clinical visit-PROactive Physical Activity in COPD (C-PPAC) questionnaire will be used to generate scores for amount of physical activity, difficulty with physical activity and total physical activity experience. C-PPAC scores will be calculated by combining questionnaire items with two variables from activity monitors (steps/day and vector magnitude units (VMU)/min). Scores range from 0 to 100, where higher numbers indicate a better score. The minimum clinically important difference (MCID) is 6 for the amount and difficulty scores and 4 for the total score.
Change in Pulmonary Rehabilitation Adapted Index of Self-Efficacy | 52 weeks
  The Pulmonary Rehabilitation Adapted Index of Self-Efficacy (PRAISE) tool is a 15-item disease-specific questionnaire that measures pulmonary rehabilitation-specific self-efficacy. The score ranges from 15 to 60, with higher scores indicating high levels of self-efficacy. The minimum clinically important difference (MCID) is 1.5 units.
Change in Pittsburgh Sleep Quality Index | 52 weeks
  The Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality over a 1-month time interval. It has 7 components (sleep quality, latency, duration, efficiency, disturbance, medication use, and daytime dysfunction) that are each scored from 0 to 3 for a total PSQI score of 0 to 21, with higher scores indicating worse sleep quality. The minimum clinically important difference (MCID) is 3 units.
Change in Hospital Anxiety and Depression Scale | 52 weeks
  The Hospital Anxiety and Depression Scale (HADS) will be used to measure symptoms of anxiety and depression. The HADS contains 14 items and consists of two subscales: anxiety and depression. Each item is rated on a four-point scale, with maximum scores of 21 for anxiety and depression. The minimum clinically important difference (MCID) is 1.5 units.
Change in The modified Medical Research Council score | 52 weeks
  The modified Medical Research Council (mMRC) has 5 questions that assess dyspnea in a graded fashion and quantify symptoms in COPD. The minimum clinically important difference (MCID) is 0.7.
Change in St. George's Respiratory Questionnaire | 52 weeks
  The St. George's Respiratory Questionnaire (SGRQ) is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. It consists of 40 questions, and scores range from 0 to 100, with higher scores indicating worse quality of life. The minimum clinically important difference (MCID) is 4 units.
Change in six-minute walk distance | 52 weeks
  The six-minute walk test is an assessment of functional capacity, and is the distance walked in 6 minutes. The minimum clinically important difference (MCID) for COPD is 26 m.
Change in University of California, San Diego Shortness of Breath Questionnaire score | 52 weeks
  The University of California, San Diego Shortness of Breath Questionnaire (SOBQ) is a 24-question, self-administered questionnaire which rates dyspnea associated with activities of daily living. Scores range from 0 to 120, with higher scores indicating greater dyspnea. The minimum clinically important difference (MCID) is 5.
All-cause mortality | 52 weeks
  Any mortality will be recorded for the 52 weeks after index hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Surya P Bhatt, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - University of Maryland, College Park, Maryland
  - Boston VA Hospital, Boston, Massachusetts
  - HealthPartners Institute, Bloomington, Minnesota
  - Minnesota VA HealthCare System, Minneapolis, Minnesota
  - Northern Westchester Hospital/Northwell Health, Chappaqua, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - Cincinnati VA Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared through a password-protected website maintained without cost to researchers after requests are vetted by the principal investigators at UAB. The investigators will make the data and associated documentation available to users under a data sharing agreement that accounts for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Users must also agree to the conditions of use governing access to the public release of data, reporting responsibilities, restrictions on redistribution of the data to third parties, and proper acknowledgement of the data resource. Research data will be de-identified to prevent disclosure of personal identifiers and presented in a summary format.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available 12 months after study completion.
Access Criteria: With approval from the Publications and Presentations Committee